CLINICAL TRIAL: NCT01899794
Title: Efficacy of a Combined Surgical and Pharmacological Therapy to Treat Mixed Urinary Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Ottawa General hospital, Ottawa University, Ottawa, Ontario, Canada (Unknown)
Responsible Party: Principal Investigator, Jacques Corcos, Professor of Urology, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-008
Record Dates: First submitted 2013-07-08; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Urinary Incontinence Mixed (Stress and Urge)
MeSH Terms: interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TVT-O (Active Comparator): mid-urethral sling
  Interventions: Procedure: TVT-O/Oxytrol; Drug: Oxytrol
- Oxytrol (Active Comparator): medication
  Interventions: Procedure: TVT-O/Oxytrol; Device: TVT-O

INTERVENTIONS:
Procedure: TVT-O/Oxytrol
  Other Names: TVT-O; Oxytrol-TDS
Device: TVT-O
  Arms: Oxytrol
Drug: Oxytrol
  Arms: TVT-O

SUMMARY:
The purpose of this study is to determine in female patients who suffer mixed urinary incontinence (MUI) the following: 1) the proportion of patients that are cured or improved by a single modality therapy (drug or surgery alone), cured or improved by a combined therapy (drug and surgery in any order) or non-responders to any of theses therapies; 2) which of the combined therapy sequences (surgery first, then followed by oral drug therapy or oral drug therapy first, then followed by surgery) is the most effective in patients needing combined therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
2. Female outpatients older than 18 years.
3. Naïve* mixed urinary incontinence (MUI) consisting of involuntary urine leakage associated with urge incontinence and incontinence with physical exertion, coughing, sneezing, etc.
4. Positive Cough Stress Test (CST):

   A positive CST is confirmed with visualization of urine leakage at the external urethral opening, concurrent with a vigorous cough and following filling of the bladder at capacity
5. Positive 24-hours Pad Test (PT):

   A positive SPT is confirmed with leakage of >8.0g/24h of urine into a pad placed over the external urethral opening. After 24 hours the pads are placed in the sealable plastic, which is weighed and the urine lost during the 24-h period is calculated
6. Daytime voiding frequency equal to or greater than to 8 times per day, with night time frequency > to 2 times per night.
7. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, the self-completion of study questionnaires and diary, and other trial procedures.
8. Urgency or urge incontinence defined by a score at the overactive bladder symptom score (OABSS) > 25 and/or urodynamic signature of the urge incontinence consisting in any uninhibited detrusor contraction during the filling phase of the CMG.

   * Naïve MUI means that the patient never received Oxytrol (oxybutynin) or surgical treatment for this condition.

Exclusion Criteria:

1. Symptoms of MUI < 6 months.
2. History of uncontrolled narrow angle glaucoma.
3. History of relevant neurological disease (e.g. multiple sclerosis).
4. History of lower urinary tract anatomical anomaly, e.g., grades 2 to 4 urogenital prolapse (at or beyond the hymen with valsalva).
5. History or evidence of urinary outlet obstruction or urinary retention, including post void residual (PVR) urine volume > 50ml
6. Chronic persistent local pathology that may cause urinary symptoms, e.g. interstitial cystitis, tumour, bladder stone.
7. Subjects using any pharmacological agent or device for their urinary incontinence less than 6 weeks prior to the inclusion or having ever used Oxytrol (oxybutynin)
8. Subjects with any of the following conditions:

   1. Indwelling urinary catheters or who perform Intermittent Self Catheterization (ISC)
   2. Passive urinary incontinence (e.g., vesico-vaginal fistula).
   3. Not capable of independent toileting.
9. Subjects with a documented and untreated UTI (temporary exclusion)
10. Subjects who require Hormone Replacement Therapy (HRT) must have been taking this at a stable dose for at least 3 months prior to study entry. Any change in dose or type of HRT taken during the study will be considered a protocol violation.
11. Subjects who are pregnant or lactating.
12. Subjects with uncontrolled narrow angle glaucoma (opinion of treating ophthalmologist will be required).
13. Subjects who have; on urodynamic investigation evidence of a poor bladder compliance and/or neurogenic detrusor hyperactivity.
14. Subjects who in the opinion of the investigator or that of the trial Clinician, are unable and/or unlikely to comprehend the nature, scope and possible consequences of the study and to follow the study procedures and instructions and complete all study related measurements. This includes poor compliance with the trial medication, and subjects who demonstrate uncooperative behaviour.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Urinary continence (measured by weighed 24-h Pad test) | 12 weeks
  Cure is defined by a 24-h pad-test of ≤ 8 g

SECONDARY OUTCOMES:
3-day urinary diary | 12 weeks
  number of leaks per day, number of pads per day,number and volume of micturitions per day

OTHER OUTCOMES:
Changes in QoL (IIQ-7 and ICIQ-SF questionnaires) and satisfaction measured by Likert scale | 12 weeks
Safety outcomes | 12 and 56 weeks
  Physical examination findings, incidence of adverse effects (AEs) and complications(erythema,pruritus,dry mouth,constipation,headache acute urinary retention,perineal pain,UTI) and PVR volume measurements (by ultrasonography)